CLINICAL TRIAL: NCT03908931
Title: Descriptive Study of the Reconstruction of Osteochondral Lesions of the Knee: Clinical and Imaging Results
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Nicolas Pujol, Principal Investigator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P19/02
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Osteochondral Defect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI (Experimental)
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: MRI — Follow up of osteochondral surgery by MRI and clinical examination

SUMMARY:
The purpose of this study is to evaluate the clinical results and MRI imaging of autologous cartilage reconstructions or collagen matrix of the knee.

There is currently little data in the literature on clinical outcomes and imaging of this type of lesion.

ELIGIBILITY:
Inclusion Criteria:

* cartilaginous reconstruction by autologous transplant or collagenous chondro-inducing knee matrix
* > 18 years

Exclusion Criteria:

* Other cartilaginous reconstruction techniques,
* other than knee joint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative knee function assessed by clinical examination | 2 years post surgery
Postoperative knee function assessed by scores | 2 years post surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CH de Versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No